CLINICAL TRIAL: NCT05018676
Title: A Single-arm, Single-center Phase II Clinical Study of Recombinant Humanized Anti-HER2 Monoclonal Antibody-AS269 Conjugate (ARX788) in the Treatment of Unresectable and/or Metastatic Breast Cancer With Low Expression of HER2
Brief Title: ARX788 in Breast Cancer With Low Expression of HER2
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xichun Hu, Professor, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACE-Breast-07
Record Dates: First submitted 2021-08-22; First posted 2021-08-24 (Actual); Last update posted 2022-04-25 (Actual); Status verified 2022-04

CONDITIONS: Breast Cancer With Low Expression of HER2
Keywords: ARX788; Breast cancer; Low expression of HER2
MeSH Terms: conditions — Breast Neoplasms | interventions — ARX788

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ARX788 (Experimental)
  Interventions: Drug: ARX788

INTERVENTIONS:
Drug: ARX788 — 1.5 mgkg IV infusion on Day 1 of each 21-day treatment cycle.

SUMMARY:
A Phase 2 Study of ARX788 in unresectable and/or metastatic breast cancer with low expression of HER2.

DETAILED DESCRIPTION:
A single arm, phase 2 study of ARX788 in unresectable and/or metastatic breast cancer with low expression of HER2. Subjects should received ≥2 lines of systemic chemotherapy regimens for recurrent or metastatic disease, and for HR positive subjects, also need to have received ≥2-line endocrine therapy ± targeted therapy (including neoadjuvant/adjuvant therapy). HER2 low expression is defined as HER2 IHC 1+ or HER2 IHC 2+ and FISH negative. The ARX788 will be administered every 3 weeks (Q3W) intravenous (IV) infusion.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to understand and sign an informed consent inform;
* Age ≥18 years, and ≤75 years, male or female;
* Diagnosed as HR arbitrary/HER2 low expression unresectable and/or metastatic breast cancer. HER2 low expression is defined as HER2 IHC 1+ (FISH negative or FISH not done) or HER2 IHC 2+ and FISH negative;
* Received ≥2 lines of systemic chemotherapy regimens for recurrent or metastatic disease, and for HR positive subjects, also need to have received ≥2-line endocrine therapy ± targeted therapy (including neoadjuvant/adjuvant therapy);
* Never had a HER2 positive result (IHC 3+ or FISH+) in previous pathological examinations;
* Have archived or fresh tumor tissue samples for HER2 status confirmation;
* According to the RECIST 1.1 standard, there is at least one measurable lesion;
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or1; LVEF≥50%;
* Adequate organ functions;
* Acute toxicities from any prior therapy, surgery, or radiotherapy must have resolved to Grade ≤1;
* Life expectancy ≥ 3 months.

Exclusion Criteria:

* History of allergic reactions to any component of ARX788, or with a history of protein drug allergy, a history of specific allergies (asthma, rheumatism, eczematous dermatitis), or a history of other severe allergic reactions, who are unsuitable for ARX788 treatment as per the investigator's judgments;
* Previous treatment with T-DM1 or other HER2-ADC drugs;
* Have other malignant tumors within 5 years before signing the informed consent form (except for non-melanoma skin cancer, cervical carcinoma in situ or other tumors that have been effectively treated, except malignant tumors that are considered cured);
* Have primary central nervous system (CNS) tumors or CNS metastases;
* Prior history of interstitial pulmonary disease requiring hormone therapy, drug-induced interstitial pulmonary disease, radiation pneumonia, or current clinically active interstitial pulmonary disease;
* Suffering from keratitis, corneal diseases, retinal diseases or active eye infections that require intervention;
* Unwilling or unable to stop wearing contact lenses for the duration of the study;
* Cardiac insufficiency;
* Uncontrolled hypertension;
* Suffering severe or uncontrolled systemic diseases;
* Had chemotherapy, radiotherapy, or immunotherapy within 4 weeks before the first dose;
* Had breast cancer endocrine therapy within 2 weeks before the first dose;
* Had palliative radiotherapy for bone metastasis within 2 weeks before the first dose;
* Any uncontrolled infection, or other conditions that may limit trial compliance or interfere with evaluation;
* Current known active infection with human immunodeficiency virus (HIV), hepatitis B virus, hepatitis C virus or syphilis;
* Plan to receive major surgical treatment within 2 weeks before first dose or during the trial period, or have suffered severe traumatic injury;
* Pregnancy or lactation;
* Unwilling or unable to use acceptable methods for contraception during the entire treatment period of this trial and within 8 months after the last dose;
* Participated in other clinical trials and used other experimental drugs within 4 weeks before the first dose;
* Any mental or cognitive impairment may limit their understanding and implementation of the informed consent form;
* Not suitable for participating in this trial, such as poor compliance.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Objective remission rate (ORR) | 2 years
  ORR is defined as the percentage of subjects who have achieved complete response and partial response according RECIST 1.1

SECONDARY OUTCOMES:
Progression-free survival (PFS) | 2 years
  PFS is defined as the time between date of first dose of study therapy and date of progression or death, whichever occurs first, will be computed for response evaluable subjects. Subjects will be censored at time of subsequent therapy
Overall survival (OS) | 2 years
  Overall survival (OS) is defined as the time from first dose of study therapy to the date of death (any cause). Subjects who are alive will be censored at the last known time that the subject was alive
Disease control rate (DCR) | 2 years
  Disease control rate (DCR) is defined as cases where objective remission (assessed as complete remission or partial remission according to RECIST 1.1 standard) or stable disease during the study
Duration of relief (DOR) | 2 years
  DOR is defined as the time from the first documented objective response (CR or PR) to the first documented disease progression or death

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No